CLINICAL TRIAL: NCT05782192
Title: A Multi-center, Randomized, Double-blind, Placebo/Positive Parallel Phase III Clinical Trial to Evaluate the Efficacy and Safety of SAL067 in Type 2 Diabetes Patients Who Cannot Effectively Control Blood Glucose Through Diet and Exercise
Brief Title: SAL067 Treatment in Patients With Type 2 Diabetes Who Are Not Controlled With Diet and Exercise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAL067-C-009; CTR20192469 (Other: NMPA); ChiCTR2000034343 (Other: Chinese Clinical Trial Registry)
Record Dates: First submitted 2023-03-09; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SAL067 (Experimental): SAL067 12mg once daily
  Interventions: Drug: SAL067
- Alogliptin (Active Comparator): Alogliptin 25mg once daily
  Interventions: Drug: Alogliptin
- placebo (Placebo Comparator): placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAL067 — SAL067 6mg(2 tablet) and placebo 25mg (1 tablet)
  Other Names: SAL067 Group
  Arms: SAL067
Drug: Alogliptin — Alogliptin 25mg(1 tablet) and placebo 6mg (2 tablet)
  Other Names: Alogliptin Group
  Arms: Alogliptin
Drug: Placebo — placebo 6mg (2 tablet) and placebo 25mg (1 tablet)
  Other Names: Placebo Group
  Arms: placebo

SUMMARY:
This is the first phase 3 randomized, double-blind, placebo/active-controlled clinical study to evaluate the efficacy and long-term safety of SAL067 in treatment-naive T2DM patients uncontrolled with diet and exercise intervention, comprising 24 weeks of double-blind treatment period followed by an open-label treatment period, making up a total of 52 weeks.

DETAILED DESCRIPTION:
All eligible subjects would enter the 24 weeks of double-blind treatment period and were randomized into the SAL067 group (12 mg once daily) or alogliptin group (25 mg once daily) or placebo group at a 2:1:1 ratio. After 24 weeks of double-blind treatment, subjects would enter the extended open-label treatment period. Subjects in the placebo group were to be switched to SAL067 (12 mg once daily) treatment, while patients in the SAL067 and alogliptin groups continued the same treatment until the end of the whole 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes patients who meet the diagnostic criteria for diabetes issued by the World Health Organization (WHO) in 1999;
2. Men or women aged 18 to 75 years old at the day of signing the informed consent;
3. Body mass index: BMI 19kg/m2 to 35kg/m2, [BMI=weight (kg)/height 2 (m2)];
4. Glycated hemoglobin (HbA1c): Screening period: HbA1c 7.5% to 10.5% (tested by the research center), when randomly enrolled: HbA1c 7.0% to 10.0% (central laboratory test) Measurement);
5. Screening period and random time fasting blood glucose <=13.9mmol/L;

Exclusion Criteria:

1. Drug compliance during the introduction period <80% or >120%;
2. Use other hypoglycemic drugs other than test drugs during the introduction period;
3. The patient may have any contraindications, allergies or hypersensitivity to fuglitagliptin (including study drug and placebo) or its excipients, DPP4 drugs, metformin;
4. Before screening, have any of the following endocrine-related medical history or evidence:

   * Diabetes other than type 2 diabetes, such as type 1 diabetes, single-gene mutation diabetes, diabetes caused by pancreatic injury or secondary diabetes, such as diabetes caused by Cushing's syndrome or acromegaly;
   * diabetic ketoacidosis, hyperglycemia and hyperosmolarity, lactic acidosis and other acute complications of diabetes within 6 months before screening;
   * severe hypoglycemia episodes (such as sleepiness caused by hypoglycemia, unconsciousness, nonsense, and even coma), or a serious history of unconscious hypoglycemia;
5. Before screening, there is a history or evidence of any of the following diseases:

   * Unstable angina, stroke or transient ischemic attack, myocardial infarction, coronary artery bypass graft or percutaneous coronary intervention (diagnostic angiography is allowed of);
   * Decompensated heart failure before screening (New York Heart Association NYHA heart function grades III and IV, persistent and clinically significant arrhythmia;
   * A history of acute and chronic pancreatitis, symptomatic gallbladder disease or history of pancreatic injury, etc. may lead to high risk factors for pancreatitis;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 458 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
HbA1c change from baseline at week 24 | Baseline and week 24
  Change From Baseline in Hemoglobin A1c (HbA1c) at week 24

SECONDARY OUTCOMES:
HbA1c change from baseline at week 4、week 12、week 40 and week 52 | Baseline 、week 4、week 12、week 40 and week 52
  Change From Baseline in Hemoglobin A1c (HbA1c) at week 4、week 12、week 40 and week 52
FPG change from baseline at week 4、week 8、week 12、week16、week24、week 40 and week 52 | Baseline、week 4、week 8、week 12、week16、week24、week 40 and week 52
Percentage of patients with HbA1c <7.0% and HbA1c <6.5% at week 24 and week 52 | Baseline 、week 24 and week 52
Percentage of patients required use of rescue therapy at week 24 and week 52 | Baseline 、week 24 and week 52
Fasting c-peptide change from baseline at week 24 and week 52 | Baseline 、week 24 and week 52
Insulin sensitivity change (calculated by HOMA-IS) from baseline at week 24 and week 52 | Baseline 、week 24 and week 52
Pancreatic β-cell function change (calculated by HOMA-β ) from baseline at week 24 and week 52 | Baseline 、week 24 and week 52

CONTACTS AND LOCATIONS:
Overall Officials: Li Yan, Ph.D, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- 1. Sun Yat-sen Memorial Hospital, Sun Yat-sen University,, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu M, Sun K, Xu W, Wang C, Yan D, Li S, Cong L, Pi Y, Song W, Sun Q, Xiao R, Peng W, Wang J, Peng H, Zhang Y, Duan P, Zhang M, Liu J, Huang Q, Li X, Bao Y, Zeng T, Wang K, Qin L, Wu C, Deng C, Huang C, Yan S, Zhang W, Li M, Sun L, Wang Y, Li H, Wang G, Pang S, Zheng X, Wang H, Wang F, Su X, Ma Y, Zhang W, Li Z, Xie Z, Xu N, Ni L, Zhang L, Deng X, Pan T, Dong Q, Wu X, Shen X, Zhang X, Zou Q, Jiang C, Xi J, Ma J, Sun J, Yan L. Fotagliptin monotherapy with alogliptin as an active comparator in patients with uncontrolled type 2 diabetes mellitus: a randomized, multicenter, double-blind, placebo-controlled, phase 3 trial. BMC Med. 2023 Oct 9;21(1):388. doi: 10.1186/s12916-023-03089-x. PMID 37814306